CLINICAL TRIAL: NCT06832072
Title: Mixed Reality Versus Manikin Simulation in Basic Life Support Training for Medical Students: a Noninferiority Randomized Controlled Trial.
Brief Title: MIxed ReAlity Versus Manikin Simulation in Basic Life Support Training for Medical Students: a Noninferiority Randomized Controlled Trial (MIRA).
Acronym: MIRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sorbonne University (Other)
Responsible Party: Principal Investigator, Anne-Laure Philippon, Principal Investigator, Sorbonne University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CER-2023-ART-SIM
Record Dates: First submitted 2025-02-07; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Medical Education; Simulation-based Methodology; Virtual Reality; Cardiac Arrest (CA); Medical Students
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MR-BLS (Experimental): Control group. In MK, medical students attended a two-hour course. Each course included a 30-minute theoretical lecture on BLS steps followed by several BLS simulation scenarios using low-fidelity manikin. Each scenario was debriefed and a tablet (Laerdal Simpad®, Laerdal, Stavanger, Norway) was used to provide feedback on chest compression rate and depth. Two to three students participated together in one scenario. The teacher-to-student ratio ranged between 1:16 and 1:20.
  Interventions: Other: MR-BLS
- MK (No Intervention): Control group. In MK, medical students attended a two-hour course. Each course included a 30-minute theoretical lecture on BLS steps followed by several BLS simulation scenarios using low-fidelity manikin. Each scenario was debriefed and a tablet (Laerdal Simpad®, Laerdal, Stavanger, Norway) was used to provide feedback on chest compression rate and depth. Two to three students participated together in one scenario. The teacher-to-student ratio ranged between 1:16 and 1:20.

INTERVENTIONS:
Other: MR-BLS — In MR group, students attended a 32 minutes course, in groups of four students with one teacher. The course included 22 minutes of individual MR training using headset (HTC Vive Focus 3®) and 10 minutes of debriefing. The individual MR training contained a step-by-step BLS reminder, including chest compression practice. Then, students engaged in a standardized virtual scenario where they interacted with both virtual characters and a physical manikin torso. The headset overlaid digital elements onto the real world, allowing the students to perform BLS while receiving real-time feedback. The feedback system provided visual cues indicating whether their chest compression rate and depth were correct. The teacher-to-student ratio was 1:4
  Other Names: Medical education Device
  Arms: MR-BLS

SUMMARY:
Purpose: To compare the effectiveness of mixed reality and traditional manikin-based simulation in basic life support (BLS) training, making the hypothesis that mixed reality was non-inferior to manikin-based simulation.

Methods: Non-inferiority randomized controlled trial. Third-year medical students were randomized in two groups. The mixed reality group (MR) received 32 minutes of individual training using a virtual reality headset and a torso for chest compressions (CC). The manikin simulation group (MK) participated in 2 hours of group training with theoretical and practical sessions using a low-fidelity manikin. The primary outcome was the overall BLS performance score, assessed at one month through a standardized BLS scenario, using a 10-item assessment scale. The quality of CC, students' satisfaction and confidence levels were secondary outcomes, assessed through superiority analyses.

DETAILED DESCRIPTION:
1.A. Context and Scientific Rationale

Out-of-hospital cardiac arrest is associated with a survival rate of less than 10% after hospital discharge (1). It is well established that the early initiation of basic cardiopulmonary resuscitation (CPR) directly influences patient survival (2). Training in basic CPR is therefore essential, particularly for medical students who will be confronted with cardiac arrest situations throughout their education and professional careers.

Simulation is currently the most widely used training tool for teaching CPR. It allows for the replication of real-world conditions by using mannequins and scenarios, placing learners in a "semi-authentic" context. This enables them to practice external chest compressions (ECC), organize basic CPR by calling for help, initiating ECC, and using an automated external defibrillator (AED). Simulation has demonstrated its effectiveness in teaching both technical skills and non-technical skills such as teamwork and communication (3,4).

New teaching methods, such as augmented reality (AR), allow immersion in virtual scenarios and interaction between physical and digital elements (5). Students can perform ECC on a mannequin while being immersed in a virtual scenario. Evaluating these new technologies is relevant to identify devices that could improve or innovate basic CPR training.

1.A.1. Current Practices in Basic CPR Training

Current training programs integrate various steps of the survival chain according to the European Resuscitation Council (ERC) guidelines (6). These steps include early recognition of cardiac arrest, calling emergency services, initiating chest compressions, and using an AED. Health simulation provides an immersive approach, exposing learners to simulated cardiac arrest situations with varying levels of realism. Using simulation mannequins, students can practice chest compressions and coordinate different CPR steps. Scenarios can be adapted to reflect different contexts, from hospital settings to emergency situations in daily life. This pedagogical approach enhances skill retention and builds confidence in responding effectively to emergencies (3). Furthermore, simulation offers a risk-free environment where errors can be identified and corrected, reinforcing hands-on learning.

1.A.2. Evaluating the Use of Virtual and Augmented Reality in Basic CPR Training

A scoping review of the literature (Dubreucq et al., in submission) was conducted to assess the use of virtual and augmented reality in basic CPR training. The analysis of 22 included studies did not conclude that virtual or augmented reality training was superior to "traditional" training, as control groups varied greatly across studies, making comparisons difficult. The primary assessment criteria used included theoretical knowledge, overall CPR performance, and the quality of ECC. The latter parameter is the most frequently evaluated and appears to be relevant due to its direct impact on survival (7).

1.A.3. Study Objectives

The present study aims to compare two CPR teaching methods: one using an augmented reality device and the other employing conventional simulation-based training. The quality of CPR performed by participants in both groups will be compared after training.

1. B. Objectives and Hypotheses

   This is a single-blind, non-inferiority randomized controlled trial comparing basic CPR training using augmented reality (AR group) to low-fidelity simulation-based training, which is currently used at the medical school (control group).

   The primary objective is to compare the overall CPR performance of both groups in a 2-minute scenario, assessed one month after training using a 10-item checklist (Appendix 1).

   Secondary objectives will be detailed afterward.

   General Hypothesis

   The study hypothesis is that augmented reality is at least as effective as low-fidelity simulation for learning basic CPR.
2. MATERIALS AND METHODS

2.A. Participants

Number of Participants: 225

Recruitment Method:

Third-year medical students at Sorbonne University participating in the mandatory "Cardiac Arrest Level 1" training.

All students enrolled in the training will receive an email with an information notice and will be invited to sign a consent form after attending a preliminary information session explaining the study.

Participation in the study is independent of participation in the mandatory training; students may decline to participate and will still attend the regular training session using traditional mannequin-based simulation.

The one-month assessment will be presented as optional for study participants, who may withdraw at any time.

Inclusion Criteria: Third-year medical students attending "Cardiac Arrest Level 1" training.

Exclusion Criteria: Declining participation in the study, physical inability to perform basic CPR (self-reported).

Randomization: After consent is obtained, participants will be randomized by training date. Sessions will be assigned randomly to the "simulation" or "augmented reality" group, with 16 students per AR session and 16-20 students per simulation session. Randomization will occur one month before the start of training. Non-participating students will attend standard simulation training without randomization.

ELIGIBILITY:
Inclusion Criteria:

* 3rd year medical students
* engaged in a universitary course "cardiac arrest"

Exclusion Criteria:

* refusal to participate
* incapacity to realise BLS

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Participants' overall BLS performance at one month after the course | One month after the inclusion
  Primary outcome was measured one month after the BLS course by an independent and blinded evaluator using the BLS performance score. It is a 10-item assessment scale, based on the validated Cardiff score, modified according to the 2021 ERC recommendations. It contains the BLS steps, following the chain of survival. Each item is scored as achieved (1) or not achieved (0), for a total score out of 10 points. Each student's performance was assessed through a standardized simulated cardiac arrest scenario. The evaluation followed a standardized protocol and was reported in an electronic Case Report Form (eCRF) using Google Forms©.

SECONDARY OUTCOMES:
Chest compression mean depth | One month after the inclusion
  Mean depth of chest compression , during 2 minutes of BLS
Chest compression (CC) mean rythm | One month after the inclusion
  Mean rythm of CC, during 2 minutes of BLS
Rate of optimal chest compressions (CC) | One month after the inclusion
  Rate of CC with a correct rythm (100-120/min) and with a correct depth (5-6cm)
Time to first electric shock | One month after the inclusion
  Time to first electric shock in seconds
Mixed reality tolerance | 30 minutes after the inclusion : at the end of the course.
  Look after adverse event after using mixed reality device (headache, nausaea...)
Confidence and lernears' satisfaction after the course | One month after the inclusion
  On a Likert scale : lerners report their confidence to initiate BLS, and their satisafaction regarding the course they endorsed.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Pitie-Salpetriere 83, boulevard de l'hopital, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
* study protocol
  * data of primary and secondary outcomes
  * inform consent form
Supporting Information: Study Protocol, SAP, ICF